CLINICAL TRIAL: NCT03157297
Title: Micra Atrial Tracking Using a Ventricular Accelerometer Study
Acronym: MARVEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT16064
Record Dates: First submitted 2017-05-09; First posted 2017-05-17 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Atrioventricular Conduction Block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Enrolled (Experimental): Subjects enrolled in the MARVEL study. Enrolled subjects will have the MARVEL algorithm downloaded into their implanted market released Micra device.
  Interventions: Device: MARVEL algorithm

INTERVENTIONS:
Device: MARVEL algorithm — Software download into implanted Micra device

SUMMARY:
The purpose of this study is to characterize performance of the MARVEL algorithm downloaded into the MicraTM TPS to provide atrial synchronous ventricular pacing in subjects with AV block.

A sub-study will be conducted within the Marvel study, the purpose of this study is to characterize the MARVEL algorithm in patients who were enrolled in the MARVEL study, and to collect and compare the accelerometer signals and AV synchrony at a second point in time.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been implanted with, or is expected to be implanted with a MicraTM TPS (Model MC1VR01), with remaining device longevity of 6 years or more.
* Subject is ≥ 18 years old and as per required local law.
* Subject has atrioventricular (AV) block.
* Subject (and/or witness, as applicable per local regulations) provides signed and dated authorization and/or consent per institution and local requirements.
* Subject is willing and able to comply with the protocol.

Exclusion Criteria:

* Subject is in atrial arrhythmia at the time of enrollment.
* Subject is currently enrolled or planning to participate in a potentially confounding drug or device trial during the study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.
* Subject is pregnant (if required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to MARVEL study procedures).
* Subject meets any exclusion criteria required by local law (age or other).

Additional criteria for the MARVEL Evolve Sub-study:

Inclusion criteria:

• Subjects in the MARVEL Sub-Study have previously been enrolled in the MARVEL main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Atrioventricular synchrony | Initial 24 hour period after patient enrollment
  On an individual heartbeat basis, this is defined as a right ventricular paced or sensed R-wave associated with an ECG confirmed P-wave.
MARVEL Evolve Substudy | Initial 24 hour period after patient enrollment
  Characterize the rate of atrioventricular synchrony provided by the MARVEL algorithm and compare the accelerometer signal amplitudes and the AV synchrony provided by the MARVEL algorithm with the data collected during the initial MARVEL procedure.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Baptist Hospital, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - NYU Langone Medical Center, New York, New York
- Kepler Universitätsklinikum Med Campus III, Linz, Austria
- UZ Leuven - Campus Gasthuisberg, Leuven, Belgium
- Nemocnice Na Homolce, Prague, Czech Republic, Czechia
- Odense Universitetshospital, Odense C, Denmark
- Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac, France
- Italy (2):
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Azienda Ospedaliero-Universitaria Pisana - Stabilimento di Cisanello, Pisa
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Hospital Universitari Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chinitz L, Ritter P, Khelae SK, Iacopino S, Garweg C, Grazia-Bongiorni M, Neuzil P, Johansen JB, Mont L, Gonzalez E, Sagi V, Duray GZ, Clementy N, Sheldon T, Splett V, Stromberg K, Wood N, Steinwender C. Accelerometer-based atrioventricular synchronous pacing with a ventricular leadless pacemaker: Results from the Micra atrioventricular feasibility studies. Heart Rhythm. 2018 Sep;15(9):1363-1371. doi: 10.1016/j.hrthm.2018.05.004. Epub 2018 May 11. PMID 29758405